CLINICAL TRIAL: NCT01793103
Title: Brigham and Women's Rheumatoid Arthritis Sequential Study
Acronym: BRASS
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Crescendo Bioscience (Industry); Bristol-Myers Squibb (Industry); UCB Pharma (Industry); Sanofi (Industry); Janssen, LP (Industry); Aqtual, Inc. (Industry)
Responsible Party: Principal Investigator, Nancy Shadick, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2002P0001762
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the present study is to establish a prospective observational cohort of Rheumatoid Arthritis patients in order to

1. Determine and validate biomarkers that predict drug response and toxicity in RA.
2. Determine and validate biomarkers that predict disease activity and prognosis in RA.
3. Evaluate the natural history of treated RA in terms of its clinical, functional and economic outcomes.

DETAILED DESCRIPTION:
The Registry will be a prospective observational study totaling 1600 patients diagnosed with RA. Patients who are 18 years of age or greater, are a patient at the R.B. Brigham Arthritis Center and have been diagnosed with RA meet entry criteria.

Once patients have agreed to participate and sign an informed consent form, they will undergo a detailed baseline examination to include demographic and clinical information, functional status, disease activity, comorbidity, laboratory testing and hand radiographs. RA criteria will be determined by the rheumatologist documenting ACR criteria and a medical record review. The primary outcomes of interest will be the presence of erosive and extra-articular disease, decline in functional status and significant drug toxicity. A sample of blood and urine will be stored for DNA/RNA testing. During this time either through interview or self-administered questionnaires, they will be asked information about their disease severity, functional status, resource utilization, level of fatigue, employment status, medications and adverse events. Information will be obtained at the time of enrollment in the Registry, during annual examinations, from semi-annual questionnaires and annual follow-up visits, as well as from medical records. Subjects will be followed for 5 years at which time they will be asked if they would like to consent to an additional 5 years. At the 10 year visit, subjects still enrolled will be given the option to consent for an additional 5 years. Subjects will be given the option within the consent forms to agree or not to the collection of their discarded specimens to analyze cells and soluble factors such as proteins in the blood to determine how they can affect the course of rheumatoid arthritis and how it develops in different individuals.

Patients with a billing diagnosis of RA (714.0) or seronegative inflammatory arthritis (714.9) over the age of 18 years old who are enrolled in the Robert Breck Brigham Arthritis Center will be eligible for recruitment. Rheumatologists within the Division of Rheumatology, Immunology and Allergy who evaluate patients in the R.B. Brigham Arthritis Center will be asked for permission to contact patients with a tentative diagnosis of RA based upon ICD billing code. A letter describing the study, Dr. Nancy Shadick, and the primary rheumatologist will be sent to the subject 7-10 days prior to their next scheduled visit. The consent form will be included with the letter so they will have time to discuss it with family and others. In the case of non-English speaking patients, the short form consent form will be presented and an interpreter will be supplied.

A letter describing the study, signed by Dr. Shadick, the PI, and the patient's primary rheumatologist will be sent to the patient 7-10 days prior to their next scheduled visit. An informed consent document will be sent at that time for the patient to read over and to discuss with family and others. If they are interested in participating in the study, the subject will be asked to bring the informed consent document to the appointment with their rheumatologist. Either the participating rheumatologist or research coordinator trained in explaining the protocol in detail will obtain the consent. Each research coordinator that will be involved in obtaining consents will undergo a 1 hour training session with the principal investigator, Nancy A. Shadick, MD. The investigator will review the general principles, benefits and risks of genetic analysis as well as details of the study. All subjects must be able to give consent for the study themselves.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years of age or older;
2. Are a patient registered at the R.B.Brigham Arthritis Center.
3. Have, at the time of enrollment a diagnosis of RA made by a board certified rheumatologist.
4. Are able and willing to provide informed consent.

Exclusion Criteria:

* less than 18 years of age
* do not have a diagnosis of RA
* have a history of SLE or Psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years or older with Rheumatoid Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 1598 (Actual)
Dates: Start 2003-03; Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Determine and validate biomarkers that predict drug response and toxicity in RA. | 15 years
  Determine and validate biomarkers that predict drug response and toxicity in RA.

SECONDARY OUTCOMES:
Determine and validate biomarkers that predict disease activity and prognosis in RA. | 15 years
  Determine and validate biomarkers that predict disease activity and prognosis in RA.
Evaluate the natural history of treated RA in terms of its clinical, functional and economic outcomes. | 15 years
  Evaluate the natural history of treated RA in terms of its clinical, functional and economic outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Shadick, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Shadick N, Hagino O, Praestgaard A, Fiore S, Weinblatt M, Burmester G. Association of hemoglobin levels with radiographic progression in patients with rheumatoid arthritis: an analysis from the BRASS registry. Arthritis Res Ther. 2023 May 27;25(1):88. doi: 10.1186/s13075-023-03068-w. PMID 37237405
- [Derived] Zhuo J, Xia Q, Sharma N, Gao S, Lama S, Cui J, Feathers V, Shadick N, Weinblatt ME. The Role of Shared Epitope in Rheumatoid Arthritis Prognosis in Relation to Anti-Citrullinated Protein Antibody Positivity. Rheumatol Ther. 2022 Apr;9(2):637-647. doi: 10.1007/s40744-022-00427-y. Epub 2022 Feb 16. PMID 35174462
- [Derived] Shadick NA, Gerlanc NM, Frits ML, Stolshek BS, Brady BL, Iannaccone C, Collier D, Cui J, Mutebi A, Weinblatt ME. The longitudinal effect of biologic use on patient outcomes (disease activity, function, and disease severity) within a rheumatoid arthritis registry. Clin Rheumatol. 2019 Nov;38(11):3081-3092. doi: 10.1007/s10067-019-04649-4. Epub 2019 Jul 29. PMID 31353421
- [Derived] Alemao E, Iannaccone CK, Weinblatt ME, Shadick NA. Association of Changes in Anticitrullinated Protein Antibody Levels With Resource Use and Disease Activity Measures in Rheumatoid Arthritis Patients a US Observational Cohort. Clin Ther. 2019 Jun;41(6):1057-1065.e3. doi: 10.1016/j.clinthera.2019.04.029. Epub 2019 May 23. PMID 31130229
- [Derived] Ahmad HA, Alemao E, Guo Z, Iannaccone CK, Frits ML, Weinblatt M, Shadick NA. Association of Low Bone Mineral Density with Anti-Citrullinated Protein Antibody Positivity and Disease Activity in Established Rheumatoid Arthritis: Findings from a US Observational Cohort. Adv Ther. 2018 Feb;35(2):232-242. doi: 10.1007/s12325-017-0657-x. Epub 2018 Jan 25. PMID 29368271
- [Derived] Alemao E, Guo Z, Frits ML, Iannaccone CK, Shadick NA, Weinblatt ME. Association of anti-cyclic citrullinated protein antibodies, erosions, and rheumatoid factor with disease activity and work productivity: A patient registry study. Semin Arthritis Rheum. 2018 Apr;47(5):630-638. doi: 10.1016/j.semarthrit.2017.10.009. Epub 2017 Oct 13. PMID 29241640
- [Derived] Alemao E, Joo S, Kawabata H, Al MJ, Allison PD, Rutten-van Molken MP, Frits ML, Iannaccone CK, Shadick NA, Weinblatt ME. Effects of Achieving Target Measures in Rheumatoid Arthritis on Functional Status, Quality of Life, and Resource Utilization: Analysis of Clinical Practice Data. Arthritis Care Res (Hoboken). 2016 Mar;68(3):308-17. doi: 10.1002/acr.22678. PMID 26238974